











# DYNAMIC Tanzania – MedAL-mentor ancillary study Statistical Analysis Plan (SAP)

| Protocol title | Dynamic clinical decision support algorithms to manage sick children in primary health care settings in Tanzania (DYNAMIC TZ) | | |
|---|---|---|---|
| Protocol version number | 5.0 | Date | 07.09.2022 |
| Study registration number | DYNAMIC TZ: NCT05144763 - MedAL-mentor ancillary study: NCT05901155 | | |
| SAP version number | 1.0 | Date | 18.12.2023 |

| Authors | Role | Signature | Date |
|---|---|---|---|
| Alix Miauton | Conceptualisation,<br>drafted first draft, and<br>revisions | Thouse | 18.12.2023 |
| Rainer Tan | Conceptualisation, review of the first draft | R-Z | 18.12.2023 |
| Chacha Mangu | Review of the first draft | Che Vamo | 20.12.2023 |
| Lameck Luwanda | Review of the first draft | Im te | 20.12.2023 |
| Patrick Taffé | Senior statistician,<br>drafted first draft of the<br>analysis section | Man ' | 19122023 |
| Alexandra Kulinkina | Review of the first draft | Comen Hair | 18.12.2023 |
| Valérie d'Acremont | Conceptualisation, review of the first draft | ll.al | 18.12.2023 |

#### **Revision history**

| Protocol version | Updated<br>SAP version<br>no | Section number changed | Description of and reason for change | Date<br>changed |
|---|---|---|---|---|



# **Table of contents**

| 1. | ABBREVIATIONS AND GLOSSARY OF TERMS | 3 |
|------|-------------------------------------|----|
| 2. | INTRODUCTION | 4 |
| 2.1. | | 4 |
| 2.2. | Research hypothesis | 4 |
| 2.3. | Study objectives | 5 |
| 3. | STUDY METHODS | 5 |
| 3.1. | Study design | 5 |
| 3.2. | Sample size | 6 |
| 3.3. | | |
| 3.4. | | |
| 3.5. | J | |
| 4. | STATISTICAL PRINCIPLES | 6 |
| 4.1. | Adherence and protocol deviations | 6 |
| 4.2. | Analysis population definitions | 7 |
| 5. | TRIAL POPULATION | 7 |
| 5.1. | Screening data | 7 |
| 5.2. | <b>5</b> , | |
| | 5.2.1. Health facility eligibility | 7 |
| | 5.2.2. HCWs eligibility | |
| | 5.2.3. Participants eligibility | |
| 5.3. | | |
| 5.4. | I I | |
| 6. | | 10 |
| 6.1. | | |
| | 6.1.1. Primary outcome | 10 |
| | 6.1.2. Secondary outcomes | |
| | 6.1.3. Exploratory outcomes | |
| 6.2. | , | |
| 6.3. | <b>5</b> | |
| 7. | REFERENCES | 13 |



## 1. Abbreviations and glossary of terms

CDSA Clinical Decision Support Algorithm

CI Confidence interval

CONSORT CONsolidated Standards Of Reporting Trials
eCDSA electronic Clinical Decision Support Algorithm

ePOCT+ Name of eCDSA (not an abbreviation)

GoT-HoMIS Government of Tanzania -Hospital Management Information System

HCW Health Care Worker

HF Health Facility

IQR Interquartile range

medAL-mentor Name of a monitoring and benchmarking tool (not an abbreviation)

mRDT malaria Rapid Diagnostic Test

MTUHA Mfuma wa Taarifa za Uendeshaji Huduma za Afya (TZ health

management information system)

STATA Statistical software package (not an abbreviation)

TZ Tanzania



#### 2. Introduction

## 2.1. Background and rationale

ePOCT+ is a pediatric electronic clinical decision support algorithm designed for healthcare workers in primary care centers in Tanzania. The objective is to improve the integrated management of acutely ill children aged 1 day to 14 years and reduce inappropriate antibiotic prescription.

Preliminary findings from the first phase of the DYNAMIC project, a cluster randomized controlled study, indicate a significant decrease in antibiotic prescription from 70% of all consultations in the control arm to 23% in HFs using ePOCT+, with similar clinical outcomes at day 7. This is consistent with what has been reported in previous studies with earlier generations of this eCDSA.<sup>1,2</sup> However, in DYNAMIC, there was considerable variation in antibiotic prescription and uptake of ePOCT+ across different HFs. In addition, other studies using different eCDSA based on Integrated Management of Childhood Illness guidelines did not show any impact on antibiotic prescription.<sup>3</sup> Therefore, it is crucial to better understand the factors promoting the uptake of eCDSAs and influencing antibiotic prescription.

During the first phase of the DYNAMIC project in intervention HFs, mentoring of HCWs was conducted with a real-time monitoring and benchmarking dashboard known as medAL-mentor, which relied on data collected through ePOCT+. The tool consists of an interactive dashboard enabling the study team to review trends in antibiotic prescription and other clinical indicators for each HF. The team provided direct feedback to HCWs on their performance, and compared it with data from other HFs. The team found that mentoring facilitated by this near real-time audit, feedback, and benchmarking dashboard had benefits and potentially contributed to the observed results.

This is consistent with several articles in the literature highlighting the positive impact of auditing and feedback to improve antibiotic stewardship in primary care, 4-7 although in other studies this positive effect was rather modest or absent. 8,9 Benchmarking in healthcare - defined as "a process of comparative evaluation and identification of the underlying causes leading to high levels of performance" 10- has also proven successful in primary care, not only in reducing antibiotic prescription but also in enhancing quality of care. 11-15 Indeed, benchmarking has been promoted for years by infectious disease societies as a component of hospital antimicrobial stewardship programs, 16 even if not always successful. 17 Of note, most of the feedback and benchmarking activities described in the literature have not been conducted in real-time but rather retrospectively, for instance on a monthly or quarterly basis. In addition, they required the intervention of an external party, whereas medAL-mentor also enables HCWs to access their results directly themselves. Finally, published initiatives have largely come from middle and high-income countries. 11 Overall, there is a lack of data and consensus regarding the impact of digital tools enabling real-time audit, benchmarking, and feedback on antibiotic prescription and quality of care.

The goal of this ancillary study is to reduce antibiotic prescription and improve quality of care for children in primary care in Tanzania using a near real-time monitoring and benchmarking dashboard (medAL-mentor), as well as feedback from the study team.

## 2.2. Research hypothesis

The null hypothesis is that there is no difference in antibiotic prescription between HFs with access to medAL-mentor and those without. The alternative hypothesis is that there is a difference between the two groups.

 $H_0: p_0=p_1$  $H_1: p_0>p_1$ 

 $p_0$ : antibiotic prescription in the control group  $p_1$ : antibiotic prescription in the intervention group



## 2.3. Study objectives

The primary objective of the study is to determine whether the provision of medAL-mentor, an online monitoring and benchmarking tool, decreases antibiotic prescription by primary care clinicians using a clinical decision support algorithm (ePOCT+) for the management of sick children.

Secondary objectives are:

- a. To assess the impact of medAL-mentor on clinicians' uptake of ePOCT+
- b. To assess the impact of medal-mentor on clinicians':
  - a. Performance of key measurements and assessment of signs by clinicians
  - b. Compliance with the recommendations related to point-of-care tests (for malaria and hemoglobin)

## 3. Study methods

## 3.1. Study design

MedAL-mentor study is an open-label, parallel cluster randomised controlled study embedded in the second phase of the DYNAMIC study in Tanzania. The intervention consists of providing direct access to medAL-mentor to the study team and to the HCWs. The study team will target calls and monitoring visits to HFs based on medAL-mentor indicators and use the dashboard to facilitate mentoring with HCWs. Since the intervention takes place at the HCW level and their practices are influenced by the context of the HF they are working in, randomization at the HF level rather than at the HCW level was chosen.

40 HFs using ePOCT+ for the first time during the second phase of the DYNAMIC project will be randomized into two groups (randomization 1:1, intervention: control).

In HFs allocated to the medAL-mentor arm, the intervention will consist of:

- Providing tablets with ePOCT+ and initial training for use by HCWs
- Initial training on antibiotic stewardship
- Access to medAL-mentor for HCWs and the study team
- Regular (at least every 2 weeks) supportive messages sent by the study team to HCWs providing feedback from medAL-mentor
- Targeted mentoring activities (via phone calls or HFs visits) provided by the study team, guided by the review of medAL-mentor

In HFs allocated to the control arm, tablets with ePOCT+ will also be provided to HCWs with initial training, but subsequent monitoring will be conducted routinely:

- Providing tablets with ePOCT+ and initial training for use by HCWs
- Initial training on antibiotic stewardship
- No access to medAL-mentor for HCWs or the study team
- At least one message sent by the study team to HCWs every two weeks, to inquire about any issues and trigger a call or site visit if needed
- At least one visit from the study team in each HF every two months.

The primary outcome measure is the antibiotic prescription rate as routinely documented by HCWs in the HFs (such as the MTUHA book or individual patient records). Secondary outcome measures are level of uptake of ePOCT+, antibiotic prescription rate as reported in medAL-reader, and other quality of care indicators (see below).



### 3.2. Sample size

The sample size was calculated to demonstrate an absolute reduction of 15% in antibiotic prescription in the intervention group, in a superiority analysis.

The intraclass correlation coefficient (ICC=0.08), the baseline antibiotic prescription (40%, in absence of medAL-mentor supervision), the cluster size (a conservative estimate of 80 patients/month/cluster, for 6 months), and the coefficient of variation for cluster sizes (0.6) were estimated from results of the first phase of the study. The duration (6 months) was chosen to consider the time required to induce change in HCWs' behavior and to evaluate their fatigue over time.

To have 80% power to detect an absolute difference of 15% of antibiotic prescription between the two arms, for a two-sided test at alpha of 0.05, we would require 13 clusters and 6240 participants per arm. Given the uncertainty in the estimation of the parameters used for the sample size calculation, the time estimated to induce change and in order to we decided to include all the available HFs, i.e. 20 clusters per arm.

#### 3.3. Randomization

All 40 HFs part of the DYNAMIC project and using ePOCT+ for the first time during the second phase of the project (i.e. 20 HFs that were in the control group during the first phase of DYNAMIC, and 20 HFs newly included for the second phase) will be included in the medALmentor study. HFs will be randomized (1:1, intervention:control) to have access to medALmentor (intervention) or routine monitoring (control). Randomization will be stratified by number of patients/week (< or > 25 children under five per week) and by access to GoT-HoMIS (the Tanzanian Health Management Information System), to ensure balance of these variables in the two arms. Where possible, the exposure will be randomized 1:1 within strata and misfits will be reallocated to strata to get as good as possible overall balance (i.e. similarity between the two arms).<sup>18</sup>

An independent statistician will perform the randomization.

#### 3.4. Timing of final analysis

Final analysis will be performed after collection of the outcome for 6 months in all 40 HFs included in the study (30 November 2023). All outcomes will be analysed collectively.

#### 3.5. Timing of outcome assessments

The primary and secondary outcomes will be assessed with data recorded by the HCW at the time of the consultation (day 0).

## 4. Statistical principles

All applicable statistical tests will be 2-sided and will be performed using a 5% significance level. All confidence intervals presented will be 95% and two-sided.

#### 4.1. Adherence and protocol deviations

Adherence to the medAL-mentor study protocol is assessed based on the percentage of : **Intervention** HFs with :

- Access to medAL-mentor for HCWs and the study team
- Regular supportive messages (at least every 2 weeks) to HCW with feedbacks from medAL-mentor



Targeted phone calls and visits based on medAL-mentor

#### Control HFs with:

- No access to medAL-mentor for HCWs and the study team
- At least one message every 3 weeks, to inquire about any issues and trigger a site visit if needed
- At least 1 visit every 10 weeks and at least 3 visits during the study period

% adherence intervention = (number HFs fulfilling intervention criteria above / total number of intervention HF)\*100.

% adherence  $_{control}$  = (number HFs fulfilling control criteria above / total number of control HF)\*100%.

Descriptive statistics on the adherence will be provided by study arm (intervention and control).

The following are pre-defined major protocol violations at HF level with a direct bearing on the primary outcome :

#### Intervention HF:

Not having access to medAL-mentor for the HCWs or the study team during the entire study period

#### Control HF:

Having access to medAL-mentor for the HCWs and/or the study team any time during the study period

## 4.2. Analysis population definitions

*Intention-to-treat analysis*: This analysis includes all consultations in HFs included in the study, regardless of whether the HCWs used ePOCT+ and had access to medAL-mentor.

*Per-protocol population*: This analysis includes only consultations in HFs included in the study and that did not experience major protocol violation during the study period.

## 5. Trial population

## 5.1. Screening data

Screening data will be presented for all children visiting participating HFs (see eligibility criteria below).

The total number of days recruiting, the total number of consultations with screened children and the total number of consultations with enrolled participants will be presented. The number of excluded participants from the primary and secondary outcomes analysis (with the number of those who did not provide consent and those without data available) will be presented. The summary will be provided overall and by HF.

## 5.2. Eligibility

#### 5.2.1. Health facility eligibility

HFs eligible for the medAL-mentor study are those included in the DYNAMIC study, and using ePOCT+ for the first time during the second phase of the DYNAMIC study:

- 20 HFs that were in the control group during the first phase of DYNAMIC
- 20HFs newly included for the second phase of the DYNAMIC study, selected purposively among HFs eligible for the first phase

(see SAP phase 1 for details on HF selection)



#### 5.2.2. HCWs eligibility

All clinicians working in sampled HFs will participate to the medAL-mentor study.

#### 5.2.3. Participants eligibility

A child is eligible for the medAL-mentor study if:

- they visit a HF included in the medAL-mentor study

#### **AND**

- they meet the following inclusion criteria and none of the following exclusion criteria:

#### **Inclusion Criteria:**

- Aged 1 day (24 hours) to 14 years (inclusive)
- Presenting for an acute medical or surgical condition

#### **Exclusion Criteria:**

- Presenting for scheduled consultation for a chronic disease (e.g. HIV, TB, NCD, malnutrition)
- Presenting for routine preventive care (e.g. growth monitoring, vitamin supplementation, deworming, vaccination).

Eligibility criteria will be assessed using the routine registry. For the primary outcome measure, all eligible participants will be included in the analysis.

For secondary and exploratory outcomes, whose measurement is based on ePOCT+ data, only participants managed with the tool will be included in the analysis. In addition, participants whose caregiver was unavailable, unable or unwilling to provide oral consent will be excluded from the analysis.



#### 5.3. Recruitement

A CONSORT flow diagram will be used to summarise the number of consultations with participants who were screened and enrolled and the number of consultations analysed for secondary and exploratory outcomes.



## 5.4. Baseline HF and patient characteristics

The following baseline cluster (HF) characteristics will be summarized by study arm:

- HF type (dispensary or health center) and region
- Access to GoT-HoMIS
- · Average number of patients under 15 seen per month by HF
- Baseline % antibiotic prescription by HF (as reported in ePOCT+) in the month before the start of the study (May 2023)



The baseline patient characteristics that will be summarized by study arm, and for the overall study include:

- Demographics: sex (number and percentage); age (median and IQR), age groups 0-2 months, 2 months 5 years, 5-14 years (number and percentage) (for all included participants)
- Medical history: Main reasons for consultation fever, respiratory, gastrointestinal, ear/nose/throat/mouth or skin complaint (number and percentage) (for participants with ePOCT+ data)
- Basic measurements: weight for age (median and IQR) (for participants with ePOCT+ data)

No formal statistical comparisons of baseline data will be performed.

## 6. Analysis

#### 6.1. Outcome definition

#### 6.1.1. Primary outcome

Percentage of children prescribed an antibiotic in the intervention group (medAL-mentor) as compared to the control group (routine monitoring)

**Outcome measure:** Number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation, over all eligible children, as reported by the HCWs in the routine registry

**Timing and method of assessment**: documented by the HCW at the end of the consultation, in the routine registry (day 0)

Analysis type: superiority

#### 6.1.2. Secondary outcomes

All secondary outcomes are compared between the intervention (medAL-mentor) and control (routine care) arms (superiority analysis).

#### a. Uptake of ePOCT+

Percentage of consultations with eligible children performed with ePOCT+

**Outcome measure:** number of consultations completed with ePOCT+, over all consultations with eligible children as reported in MTUHA books

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) and at the end of the consultation (routine registry), at day 0

Analysis type: superiority

#### b. Quality of care indicators

Percentage of children in whom key signs have been checked by HCWs

Number of children in whom each of the key signs (temperature, weight, MUAC, respiratory rate) has been checked by HCWs, over the total number of children for whom this was recommended, as reported by HCWs in ePOCT+



**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) at day 0

Analysis type: superiority

#### Percentage of children for whom appropriate diagnostic tests have been performed by HCWs

Number of children for whom each of the diagnostic tests (haemoglobin and malaria tests) has been performed by HCWs, over the total number of children for whom the diagnostic test was recommended, as reported by HCWs in ePOCT+

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) at day 0

Analysis type: superiority

#### 6.1.3. Exploratory outcomes

All exploratory outcomes are compared between the intervention (medAL-mentor) and control (routine care) arms.

#### a. Antibiotic prescription over time (longitudinal analysis)

**Outcome measure:** number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation, over all eligible children, every week of the study period, as reported by the HCWs in the routine registry

**Timing and method of assessment**: documented by the HCW at the end of the consultation (routine registry) at day 0

#### b. Antibiotic prescription in children managed with and without ePOCT+

**Outcome measure:** number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation, over all eligible children, as reported by the HCWs in the routine registry for children managed with and without ePOCT+

**Timing and method of assessment**: documented by the HCW at the end of the consultation (routine registry) at day 0

# c. Antibiotic prescription reported in ePOCT+ versus in routine data (data consistency)

**Outcome measure:** number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation systemic as reported by the HCW in ePOCT+ over number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation systemic as reported by the HCW in the routine registry

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) and at the end of the consultation (routine registry) at day 0



#### d. Completion of ePOCT+

**Outcome measure:** number of consultations completed with ePOCT+, over all consultations started with ePOCT+

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) at day 0

#### e. Appropriate case management for malaria

#### **Outcomes measure:**

- % of consultations with febrile children tested for malaria
- % of consultations with children with a positive malaria test prescribed an antimalarial
- % of consultations with children with a negative malaria test prescribed an antimalarial
- % of consultations with untested children prescribed an antimalarial

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) at day 0

#### f. Appropriate case management for acute respiratory infections

#### Outcomes measure:

- % of children with acute respiratory infection prescribed an antibiotic
- % of children with bacterial pneumonia prescribed an antibiotic
- % of children with viral pneumonia prescribed an antibiotic
- % of children with cough/common cold prescribed an antibiotic

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) at day 0

#### g. Appropriate case management for diarrhea

#### **Outcomes measure:**

- % of children with acute diarrhea prescribed zinc
- % of children with acute diarrhea prescribed an antibiotic

**Timing and method of assessment**: documented by the HCW during the consultation (medAL-reader) on day 0

#### 6.2. Analysis methods

Analyses will follow CONSORT guidelines. 19

All the analyses will be carried out using generalized linear mixed models (GLMM, more specifically the multilevel logistic regression model with fixed and random-effects) to account for the complex multi-level structure of the data (induced by the stratified cluster randomized procedure), with individuals measurements nested within HCWs, who are themselves nested within HFs, which in turn are nested within districts, and at the highest-level districts are nested



within regions.<sup>20</sup> For the primary outcome, available risk factors at the individual level will be age category, sex, and type of final diagnosis (gastro-intestinal, respiratory, skin, malaria, other). For secondary outcomes, available risk factors at the individual level will be age, sex, child presenting with fever, gastro-intestinal, respiratory, ear/nose/throat/mouth and/or skin problem. In addition, to account for the correlation between the two exposure groups induced by the stratification, all the analyses will be adjusted for the stratification factors used in the randomization and not already accounted for (i.e. attendance rate and use of GoT-HoMIS) in the multi-level structure. Finally, the analyses will be adjusted by the baseline antibiotic prescription at each HF.

A special random-effects structure will be used at the HF level to account for unmeasured heterogeneity of the intervention effect<sup>21</sup> and confounding by cluster will be dealt with by separating within- and between-cluster effects using a partitioning method. <sup>22,23</sup>

Interactions (i.e. effect modification) between covariables (at the individual level) and exposure (i.e. medAL-mentor vs control) will be introduced into the model as fixed-effects. Variable selection will be based on clinical relevance and not on statistical tests of significance; consequently, no correction for multiple testing will be applied.<sup>24</sup>

To assess the impact of the intervention at the population level (i.e. the population averaged effect), the two marginal probabilities in the exposed and unexposed children will be computed by marginalization of the estimated conditional probabilities. Eased on these marginal probabilities, the marginal relative risk and marginal risk difference will be computed. These marginal parameters quantify the average impact of the intervention in the whole population, and to assess the impact of the intervention in specific subgroups of children marginal probabilities will be also computed in the subpopulations defined by the risk factors detailed above.

## 6.3. Missing data

Missing values will not be imputed given the great complexity of multiple imputations in the context of complex multi-level structures.<sup>27</sup>

#### 7. References

- 1. Keitel K, Kagoro F, Samaka J, et al. A novel electronic algorithm using host biomarker point-of-care tests for the management of febrile illnesses in Tanzanian children (e-POCT): A randomized, controlled non-inferiority trial. *PLoS Med* 2017; **14**(10): e1002411.
- 2. Shao AF, Rambaud-Althaus C, Samaka J, et al. New Algorithm for Managing Childhood Illness Using Mobile Technology (ALMANACH): A Controlled Non-Inferiority Study on Clinical Outcome and Antibiotic Use in Tanzania. *PLoS One* 2015; **10**(7): e0132316.
- 3. Horwood C, Haskins L, Mapumulo S, et al. Electronic Integrated Management of Childhood Illness (elMCI): a randomized controlled trial to evaluate an electronic clinical decision-making support system for management of sick children in primary health care facilities in South Africa; 2023.
- 4. Gulliford MC, Juszczyk D, Prevost AT, et al. Electronically delivered interventions to reduce antibiotic prescribing for respiratory infections in primary care: cluster RCT using electronic health records and cohort study. *Health Technol Assess* 2019; **23**(11): 1-70.
- 5. Zhen L, Jin C, Xu HN. The impact of prescriptions audit and feedback for antibiotic use in rural clinics: interrupted time series with segmented regression analysis. *BMC Health Serv Res* 2018; **18**(1): 777.



- 6. Chang Y, Sangthong R, McNeil EB, Tang L, Chongsuvivatwong V. Effect of a computer network-based feedback program on antibiotic prescription rates of primary care physicians: A cluster randomized crossover-controlled trial. *J Infect Public Health* 2020; **13**(9): 1297-303.
- 7. Yang J, Cui Z, Liao X, et al. Effects of a feedback intervention on antibiotic prescription control in primary care institutions based on a Health Information System: a cluster randomized cross-over controlled trial. *J Glob Antimicrob Resist* 2023; **33**: 51-60.
- 8. Aghlmandi S, Halbeisen FS, Saccilotto R, et al. Effect of Antibiotic Prescription Audit and Feedback on Antibiotic Prescribing in Primary Care: A Randomized Clinical Trial. *JAMA Intern Med* 2023; **183**(3): 213-20.
- 9. Gerber JS, Prasad PA, Fiks AG, et al. Effect of an outpatient antimicrobial stewardship intervention on broad-spectrum antibiotic prescribing by primary care pediatricians: a randomized trial. *Jama* 2013; **309**(22): 2345-52.
- 10. Ellis J. All inclusive benchmarking. J Nurs Manag 2006; 14(5): 377-83.
- 11. Willmington C, Belardi P, Murante AM, Vainieri M. The contribution of benchmarking to quality improvement in healthcare. A systematic literature review. *BMC Health Serv Res* 2022; **22**(1): 139.
- 12. Piccoliori G, Mahlknecht A, Abuzahra ME, et al. Quality improvement in chronic care by self-audit, benchmarking and networking in general practices in South Tyrol, Italy: results from an interventional study. *Fam Pract* 2021; **38**(3): 253-8.
- 13. Hermans MP, Elisaf M, Michel G, et al. Benchmarking is associated with improved quality of care in type 2 diabetes: the OPTIMISE randomized, controlled trial. *Diabetes Care* 2013; **36**(11): 3388-95.
- 14. Meeker D, Linder JA, Fox CR, et al. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. *Jama* 2016; **315**(6): 562-70.
- 15. Wei X, Zhang Z, Walley JD, et al. Effect of a training and educational intervention for physicians and caregivers on antibiotic prescribing for upper respiratory tract infections in children at primary care facilities in rural China: a cluster-randomised controlled trial. *Lancet Glob Health* 2017; **5**(12): e1258-e67.
- 16. Dellit TH, Owens RC, McGowan JE, Jr., et al. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. *Clin Infect Dis* 2007; **44**(2): 159-77.
- 17. Marwick CA, Hossain A, Nogueira R, et al. Feedback of Antibiotic Prescribing in Primary Care (FAPPC) trial: results of a real-world cluster randomized controlled trial in Scotland, UK. *J Antimicrob Chemother* 2022; **77**(12): 3291-300.
- 18. Carril A. Dealing with Misfits in Random Treatment Assignment. *The Stata Journal* 2017; **17**(3): 652-67.
- 19. Campbell MK, Piaggio G, Elbourne DR, Altman DG. Consort 2010 statement: extension to cluster randomised trials. *Bmj* 2012; **345**: e5661.
- 20. Austin PC, Merlo J. Intermediate and advanced topics in multilevel logistic regression analysis. *Stat Med* 2017; **36**(20): 3257-77.
- 21. Omar RZ, Thompson SG. Analysis of a cluster randomized trial with binary outcome data using a multi-level model. *Stat Med* 2000; **19**(19): 2675-88.
- 22. Localio AR, Berlin JA, Have TRT. Confounding Due to Cluster in Multicenter Studies—Causes and Cures. *Health Services and Outcomes Research Methodology* 2002; **3**(3): 195-210.
- 23. Begg MD, Parides MK. Separation of individual-level and cluster-level covariate effects in regression analysis of correlated data. *Stat Med* 2003; **22**(16): 2591-602.
- 24. Savitz DA, Olshan AF. Multiple comparisons and related issues in the interpretation of epidemiologic data. *Am J Epidemiol* 1995; **142**(9): 904-8.
- 25. Miglioretti DL, Heagerty PJ. Marginal modeling of nonnested multilevel data using standard software. *Am J Epidemiol* 2007; **165**(4): 453-63.
- 26. Muff S, Held L, Keller LF. Marginal or conditional regression models for correlated non-normal data? *Methods in Ecology and Evolution* 2016; **7**(12): 1514-24.



